CLINICAL TRIAL: NCT01009814
Title: Randomized, Open Label, Multiple-Dose Study to Evaluate the Pharmacodynamics, Safety and Pharmacokinetics of BMS-663068 in HIV-1 Infected Subjects
Brief Title: Pharmacodynamics, Safety and Pharmacokinetics of BMS-663068, an HIV Attachment Inhibitor, in HIV-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206267; AI438-006 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-10

CONDITIONS: HIV Infections
Keywords: HIV, HIV attachment inhibitor, attachment inhibitor
MeSH Terms: conditions — HIV Infections | interventions — fostemsavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- BMS-663068 600 mg Q12H + RTV 100 mg Q12H (Experimental): All participants received BMS-663068 600 milligram (mg) and Ritonavir (RTV) 100 mg every 12 hours (Q12H) from Day 1 to Day 8.
  Interventions: Drug: BMS-663068; Drug: Ritonavir
- BMS-663068 1200 mg QHS + RTV 100 mg QHS (Experimental): All participants received BMS-663068 1200 mg and RTV 100 mg every night (quaque hora somni [QHS]) from Day 1 to Day 8.
  Interventions: Drug: BMS-663068; Drug: Ritonavir
- BMS-663068 1200 mg Q12H + RTV 100 mg Q12H (Experimental): All participants received BMS-663068 1200 mg and RTV 100 mg Q12H from Day 1 to Day 8.
  Interventions: Drug: BMS-663068; Drug: Ritonavir
- BMS-663068 1200 mg Q12H + RTV 100 mg QAM (Experimental): All participants received BMS-663068 1200 mg Q12H and RTV 100 mg every 24 hours in the morning (quaque ante meridiem [QAM]) from Day 1 to Day 8.
  Interventions: Drug: BMS-663068; Drug: Ritonavir
- BMS-663068 1200 mg Q12H (Experimental): All participants received BMS-663068 1200 mg Q12H from Day 1 to Day 8.
  Interventions: Drug: BMS-663068

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068 will be administered as a tablet formulation
Drug: Ritonavir — Ritonavir will be administered as a capsule.
  Arms: BMS-663068 1200 mg Q12H + RTV 100 mg Q12H; BMS-663068 1200 mg Q12H + RTV 100 mg QAM; BMS-663068 1200 mg QHS + RTV 100 mg QHS; BMS-663068 600 mg Q12H + RTV 100 mg Q12H

SUMMARY:
Research Hypothesis: Administration of BMS-663068, a prodrug for HIV attachment inhibitor BMS-626529, will result in a mean decrease of at least 1 log10 in HIV RNA at Day 9 following 8 days of therapy in at least one dosing regimen that is safe and well tolerated in Clade B HIV-1 infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Clade B HIV-1 infected subjects meeting following criteria at screening:

  * Plasma HIV RNA ≥ 5,000 copies/mL
  * CD4+ lymphocyte ≥ 200 cells/µL
  * Antiretroviral naive or experienced
  * Off all ARV therapy with HIV activity for > 8 weeks
* BMI of 18 to 35 kg/m2, inclusive.
* Not currently co-infected with HCV or HBV
* Men and women, ≥ 18 years of age

Exclusion Criteria:

* Woman of childbearing potential (WOCBP) unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period up to 12 weeks after the last dose of study drug.
* WOCBP using prohibited contraceptive method including oral, injectable, or implantable hormonal contraceptive agent within 12 weeks of enrollment.
* Women who are pregnant or breastfeeding.
* Women with positive pregnancy test on enrollment or prior to study drug intake.
* Sexually active fertile men not using effective birth control during study and for at least 12 weeks after last dose of study drug if partners are WOCBP.
* Significant acute or chronic medical illness not stable or not controlled with medication or not consistent with HIV infection.
* Current or recent (within 3 months) gastrointestinal disease that, in the opinion of Investigator or Medical Monitor, may impact on drug absorption and/or put subject at risk for GI tract irritation and/or bleeding.
* Acute diarrhea lasting ≥ 1 day, within 3 weeks prior to randomization.
* Major surgery within 4 weeks of study drug intake.
* Gastrointestinal surgery that could impact upon absorption of study drug.
* Donation of blood or plasma to blood bank or in a clinical study (except a Screening visit or follow up visit of less than 50 mL) within 4 weeks of study drug intake.
* Blood transfusion within 4 weeks of study drug intake.
* Inability to tolerate oral medication.
* Inability to be venipunctured and/or tolerate venous access.
* Personal history of clinically relevant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de pointes.
* Personal or family history of long QT syndrome.
* Recent (within 6 months) drug/alcohol abuse
* Any other medical, psychiatric and/or social reason which, in the opinion of the Investigator, would make the candidate inappropriate for participation.
* Evidence of organ dysfunction or clinically significant deviation from normal in physical examination, vital signs, ECG or clinical lab determinations or not consistent with subject's degree of HIV infection.
* Evidence of 2nd or 3rd degree heart block at screening or Day -1
* Positive urine drug screen at Screening or Day -1 without valid prescription (subjects positive for cannabinoids and/or amphetamines will be included).
* Positive blood screen for hepatitis B surface antigen.
* Positive blood screen for hepatitis C antibody and hepatitis C RNA.
* History of significant drug allergy
* Exposure to any investigational drug or placebo within 4 weeks of study drug intake.
* Prescription drugs within 4 weeks prior to study drug intake, unless approved by BMS medical monitor.
* Other drugs, including over-the-counter medications, vitamins and/or herbal preparations, within 1 week prior to study drug intake, unless approved by BMS medical monitor.
* Use of oral, injectable or implantable hormonal contraceptive agent within 12 weeks of study drug intake.
* Use of prescription drugs or OTC drugs that may cause GI tract irritation or bleeding within 2 weeks of study drug intake, unless approved by BMS medical monitor.
* Use of alcohol-containing beverages within 3 days prior to study drug intake.
* Use of grapefruit, grapefruit-containing or Seville orange-containing products within 7 days prior to study drug intake.
* Prisoners or subjects involuntarily incarcerated.
* Subjects compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11-23 (Actual); Primary Completion 2010-06-25 (Actual); Study Completion 2010-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Landry I, Zhu L, Abu Tarif M, Hruska M, Sadler BM, Pitsiu M, Joshi S, Hanna GJ, Lataillade M, Boulton DW, Bertz RJ. Model-Based Phase 3 Dose Selection for HIV-1 Attachment Inhibitor Prodrug BMS-663068 in HIV-1-Infected Patients: Population Pharmacokinetics/Pharmacodynamics of the Active Moiety, BMS-626529. Antimicrob Agents Chemother. 2016 Apr 22;60(5):2782-9. doi: 10.1128/AAC.02503-15. Print 2016 May. PMID 26902761
- [Derived] Ray N, Hwang C, Healy MD, Whitcomb J, Lataillade M, Wind-Rotolo M, Krystal M, Hanna GJ. Prediction of virological response and assessment of resistance emergence to the HIV-1 attachment inhibitor BMS-626529 during 8-day monotherapy with its prodrug BMS-663068. J Acquir Immune Defic Syndr. 2013 Sep 1;64(1):7-15. doi: 10.1097/QAI.0b013e31829726f3. PMID 23614999
- [Derived] Nettles RE, Schurmann D, Zhu L, Stonier M, Huang SP, Chang I, Chien C, Krystal M, Wind-Rotolo M, Ray N, Hanna GJ, Bertz R, Grasela D. Pharmacodynamics, safety, and pharmacokinetics of BMS-663068, an oral HIV-1 attachment inhibitor in HIV-1-infected subjects. J Infect Dis. 2012 Oct 1;206(7):1002-11. doi: 10.1093/infdis/jis432. Epub 2012 Aug 14. PMID 22896665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, open label, multiple-dose study to evaluate the pharmacodynamics, safety and pharmacokinetics of BMS-663068 in human immunodeficiency virus 1 (HIV-1) infected participants. The study was conducted at single center in Germany.
Pre-assignment Details: A total of 75 participants were screened, of which 25 were screen failure, and 50 eligible participants were enrolled into the study and were randomized.
Period: Overall Study
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Started | 10 | 10 | 10 | 10 | 10
Completed | 9 | 9 | 10 | 10 | 10
Not Completed | 1 | 1 | 0 | 0 | 0
Not completed — No longer met study criteria | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (8.29) | 40.7 (13.70) | 40.7 (6.53) | 38.4 (7.83) | 42.7 (8.42) | 40.8 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 0 | 3
  Male | 9 | 9 | 9 | 10 | 10 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 10 | 10 | 10 | 10 | 10 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Logarithm With Base 10 (Log10) Change From Baseline in Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) at Day 9
Description: The primary assessment of the antiviral activity of BMS-663068 was assessed on the log10 change from Baseline in HIV RNA to Day 9. Baseline was the last non-missing observation before first dose (Day 1 pre-dose) and change from Baseline was calculated by subtracting Baseline value from post-Baseline visit value. An analysis of covariance (ANCOVA) model correcting for Baseline HIV viral load and treatment group was used to test the differences in mean log10 decrease in HIV RNA at Day 9 between 2 regimen groups by antiretroviral treatment history (ARV [antiretroviral] naive, ARV experienced, and combined [ARV naive + ARV experienced]). For the combined group (ARV naive +ARV experienced) an additional ANCOVA was used correcting also for treatment history as an additional covariate. Only Clade B participants were included in the population.
Time Frame: Baseline and Day 9
Population: Pharmacodynamic Population. It comprised of all participants for whom pharmacodynamic measurements were available at Baseline and at least one other time.
Measure: Mean (Standard Error); unit: Log10 copies per milliliter (c/mL)
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 9 | 9 | 10 | 10 | 10
Log10 copies per milliliter (c/mL) | -1.3445 (0.07925) | -1.2532 (0.10610) | -1.2381 (0.10455) | -1.1888 (0.12938) | -0.8760 (0.22621)
Statistical Analysis 1: Comparison: BMS-663068 600 mg Q12H + RTV 100 mg Q12H vs BMS-663068 1200 mg QHS + RTV 100 mg QHS; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.6102, ANCOVA; Mean Difference (Net) = -0.1089, 90% CI 2-sided [-0.4656 to 0.2477], Standard Error of Mean 0.2120
Statistical Analysis 2: Comparison: BMS-663068 600 mg Q12H + RTV 100 mg Q12H vs BMS-663068 1200 mg Q12H + RTV 100 mg Q12H; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.5452, ANCOVA; Mean Difference (Net) = -0.1266, 90% CI 2-sided [-0.4758 to 0.2225], Standard Error of Mean 0.2076
Statistical Analysis 3: Comparison: BMS-663068 600 mg Q12H + RTV 100 mg Q12H vs BMS-663068 1200 mg Q12H + RTV 100 mg QAM; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.4178, ANCOVA; Mean Difference (Net) = -0.1682, 90% CI 2-sided [-0.5139 to 0.1775], Standard Error of Mean 0.2055
Statistical Analysis 4: Comparison: BMS-663068 600 mg Q12H + RTV 100 mg Q12H vs BMS-663068 1200 mg Q12H; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.0233, ANCOVA; Mean Difference (Net) = -0.4885, 90% CI 2-sided [-0.8375 to -0.1395], Standard Error of Mean 0.2075
Statistical Analysis 5: Comparison: BMS-663068 1200 mg QHS + RTV 100 mg QHS vs BMS-663068 1200 mg Q12H + RTV 100 mg Q12H; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.9314, ANCOVA; Mean Difference (Net) = -0.0177, 90% CI 2-sided [-0.3613 to 0.3259], Standard Error of Mean 0.2043
Statistical Analysis 6: Comparison: BMS-663068 1200 mg QHS + RTV 100 mg QHS vs BMS-663068 1200 mg Q12H + RTV 100 mg QAM; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.7734, ANCOVA; Mean Difference (Net) = -0.0592, 90% CI 2-sided [-0.4032 to 0.2847], Standard Error of Mean 0.2045
Statistical Analysis 7: Comparison: BMS-663068 1200 mg QHS + RTV 100 mg QHS vs BMS-663068 1200 mg Q12H; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.0702, ANCOVA; Mean Difference (Net) = -0.3796, 90% CI 2-sided [-0.7232 to -0.0360], Standard Error of Mean 0.2043
Statistical Analysis 8: Comparison: BMS-663068 1200 mg Q12H + RTV 100 mg Q12H vs BMS-663068 1200 mg Q12H + RTV 100 mg QAM; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.8359, ANCOVA; Mean Difference (Net) = -0.0415, 90% CI 2-sided [-0.3768 to 0.2937], Standard Error of Mean 0.1993
Statistical Analysis 9: Comparison: BMS-663068 1200 mg Q12H + RTV 100 mg Q12H vs BMS-663068 1200 mg Q12H; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.0759, ANCOVA; Mean Difference (Net) = -0.3619, 90% CI 2-sided [-0.6962 to -0.0275], Standard Error of Mean 0.1988
Statistical Analysis 10: Comparison: BMS-663068 1200 mg Q12H + RTV 100 mg QAM vs BMS-663068 1200 mg Q12H; Null hypothesis was that there was 0 difference in mean log10 decrease in HIV RNA at Day 9 between two groups; Test type: Other; p = 0.1155, ANCOVA; Mean Difference (Net) = -0.3203, 90% CI 2-sided [-0.6555 to 0.0149], Standard Error of Mean 0.1993

2. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 Positive (CD4+) Cell Count and Cluster of Differentiation 8 Positive (CD8+) Cell Count
Description: Blood samples were collected for evaluation of CD4+ and CD8+ cells at Baseline (Day 1, pre-dose), Day 8, Day 15 (Follow up) and Day 50 (study discharge). Baseline was the last non-missing observation before first dose (Day 1 pre-dose) and change from Baseline was calculated by subtracting Baseline value from post-Baseline visit value.
Time Frame: Baseline (Day 1 pre-dose), Day 8, Day 15 and Day 50
Population: Pharmacodynamic Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Error); unit: Cells per microliter (cells/μL)
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 9 | 9 | 10 | 10 | 10
Cells per microliter (cells/μL)
  CD4+, Day 8, n=9, 9, 10, 10, 10 | 114.2 (74.55) | 93.4 (25.12) | 109.8 (32.37) | 38.5 (41.61) | 32.0 (36.23)
  CD4+, Day 15, n=9, 9, 10, 10, 10 | 58.4 (92.14) | -6.1 (28.15) | 117.6 (27.67) | 44.6 (69.94) | 10.4 (23.38)
  CD4+, Day 50, n=9, 9, 10, 10, 9: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9
  CD4+, Day 50, n=9, 9, 10, 10, 9 | 22.0 (91.55) | -50.3 (18.06) | 71.1 (28.55) | -48.4 (61.21) | -19.2 (17.05)
  CD8+, Day 8, n=9, 9, 10, 10, 10 | 384.2 (164.35) | 189.0 (134.27) | 218.4 (125.65) | 114.9 (131.64) | 94.6 (152.73)
  CD8+, Day 15, n=9, 9, 10, 10, 10 | 64.8 (230.86) | -153.2 (137.18) | 85.6 (112.65) | -99.6 (159.83) | -4.4 (126.77)
  CD8+, Day 50, n=9, 9, 10, 10, 9: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9
  CD8+, Day 50, n=9, 9, 10, 10, 9 | -37.6 (161.11) | -292.4 (121.73) | 139.7 (95.00) | 6.0 (170.29) | -48.2 (140.55)

3. Secondary Outcome: Change From Baseline in Percent CD4+ Cell Count and Percent CD8+ Cell Count
Description: Blood samples were collected for evaluation of percent CD4+ and percent CD8+ cells at Baseline (Day 1, pre-dose), Day 8, Day 15 (Follow up) and Day 50 (study discharge). Baseline was the last non-missing observation before first dose (Day 1 pre-dose) and change from Baseline was calculated by subtracting Baseline visit value from post-Baseline visit value.
Time Frame: Baseline (Day 1 pre-dose), Day 8, Day 15 and Day 50
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent cells per microliter
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 9 | 9 | 10 | 10 | 10
Percent cells per microliter
  Percent CD4+, Day 8, n=9, 9, 10, 10, 10 | -1.0 (1.12) | 1.2 (0.97) | 0.6 (0.78) | 0.1 (0.72) | 1.4 (1.11)
  Percent CD4+, Day 15, n=9, 9, 10, 10, 10 | 1.6 (1.00) | 1.2 (0.64) | 1.4 (1.33) | 2.4 (1.11) | 0.9 (1.51)
  Percent CD4+, Day 50, n=9, 9, 10, 10, 9: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9
  Percent CD4+, Day 50, n=9, 9, 10, 10, 9 | 1.4 (0.84) | 1.1 (1.15) | 0.3 (0.90) | -1.7 (0.97) | 0.6 (1.45)
  Percent CD8+, Day 8, n=9, 9, 10, 10, 10 | 1.0 (0.76) | -0.4 (1.02) | 0.1 (1.06) | -0.3 (1.11) | -0.2 (1.20)
  Percent CD8+, Day 15, n=9, 9, 10, 10, 10 | -3.4 (0.73) | -2.8 (1.00) | -2.9 (1.49) | -4.0 (1.73) | -2.9 (1.16)
  Percent CD8+, Day 50, n=9, 9, 10, 10, 9: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9
  Percent CD8+, Day 50, n=9, 9, 10, 10, 9 | -2.2 (1.01) | -0.7 (1.22) | -0.9 (1.19) | 1.6 (1.52) | -2.4 (1.57)

4. Secondary Outcome: Number of Participants With Treatment Emergent Non-serious Adverse Event (Non-SAE) and Serious AE (SAE)
Description: An AE is any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. Any untoward medical occurrence resulting in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent serious outcomes were categorized as SAE. Treatment emergent adverse events (occurred after start of treatment) have been presented.Safety Population comprised of all randomized participants who used the trial medication at least once.
Time Frame: Up to 50 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Non-SAE | 8 | 5 | 9 | 8 | 9
  SAE | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Any Abnormality in Physical Examination
Description: A complete physical examination included, at a minimum, assessment of the Cardiovascular, Respiratory, Gastrointestinal and Neurological systems. A brief physical examination included, at a minimum assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). Any abnormality found by investigator during physical examination were recorded. Number of participants with any abnormality in physical examination during study have been reported.
Time Frame: Up to 50 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 1 | 0 | 2 | 1 | 1

6. Secondary Outcome: Number of Participants With Worst-case Abnormalities in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Vital signs including DBP and SBP were recorded. Normal ranges were as following: For DBP, lower limit: value <55 millimeter of mercury (mmHg) and change <-20 mmHg; upper limit: value >90 mmHg and change >20 mmHg). For SBP, lower limit: value <90 mmHg and change <-10 mmHg; upper limit: value >140 mmHg and change >10 mmHg. Number of participants with worst-case abnormalities are presented. Worst-case abnormality was defined as: (1) Below Normal: at least one post-Baseline assessment was below normal range, and no post-Baseline assessment was above normal range. (2) Above Normal: at least one post-Baseline assessment was above normal range, and no post-Baseline assessment was below normal range. (3) Within Normal: all post-Baseline assessments were within normal range. It was to be considered as 'Missing' when there were no post-Baseline assessments.
Time Frame: Up to 50 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  SBP, Above Normal | 0 | 3 | 1 | 0 | 1
  SBP, Below Normal | 0 | 0 | 0 | 0 | 0
  SBP, Within Normal | 10 | 7 | 9 | 10 | 9
  DBP, Above Normal | 0 | 0 | 0 | 0 | 0
  DBP, Below Normal | 0 | 0 | 0 | 0 | 0
  DBP, Within Normal | 10 | 10 | 10 | 10 | 10

7. Secondary Outcome: Number of Participants With Worst-case Abnormalities in Body Temperature, Respiratory Rate [RR], and Heart Rate [HR]
Description: Vital signs (body temperature, RR, and HR) were recorded. Normal range were: For HR, lower limit: 55 beats per minute (bpm) and change <-15 bpm; upper limit: >100 bpm and change >30 bpm). For temperature, lower limit: 36.0 Celsius; upper limit: >37.5 Celsius or change >1.7 Celsius). For RR, lower limit: 8 breaths per minute; upper limit: >16 breaths per minute or change >10 breaths per minute. Number of participants with worst-case abnormalities are presented. Worst-case abnormality was defined as: (1) Below Normal: at least one post-Baseline assessment was below normal range, and no post-Baseline assessment was above normal range. (2) Above Normal: at least one post-Baseline assessment was above normal range, and no post-Baseline assessment was below normal range. (3) Within Normal: all post-Baseline assessments were within normal range. It was to be considered as 'Missing' when there were no post-Baseline assessments.
Time Frame: Up to 50 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  HR, Above Normal | 0 | 0 | 0 | 0 | 0
  HR, Below Normal | 1 | 2 | 1 | 0 | 1
  HR, Within Normal | 9 | 8 | 9 | 10 | 9
  RR, Above Normal | 4 | 3 | 3 | 3 | 8
  RR, Below Normal | 0 | 0 | 0 | 0 | 0
  RR, Within Normal | 6 | 7 | 7 | 7 | 2
  Temperature, Above Normal | 0 | 0 | 0 | 0 | 0
  Temperature, Below Normal | 1 | 2 | 0 | 1 | 0
  Temperature, Within Normal | 9 | 8 | 10 | 9 | 10

8. Secondary Outcome: Number of Participants With Worst-case Abnormalities in Electrocardiogram (ECG) Parameters
Description: A 12-lead ECG was recorded during the study using an ECG machine that automatically measures ECG parameters. Normal range for ECG parameters were: PR interval (upper: 200 milliseconds [ms]); QRS (lower: 50 ms; upper: 120 ms); Corrected QT interval by Bazett formula (QTcB) (change from Baseline - increases by > 30 ms); Corrected QT interval by Fredericia formula (QTcF) (change from Baseline - increases by > 30 ms). Number of participants with worst-case abnormalities are presented which was defined as: (1) Below Normal: at least one post-Baseline assessment was below normal range, and no post-Baseline assessment was above normal range. (2) Above Normal: at least one post-Baseline assessment was above normal range, and no post-Baseline assessment was below normal range. Within Normal: all post-Baseline assessments were within normal range. It was to be considered as 'Missing' when there were no post-Baseline assessments.
Time Frame: Up to 50 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  PR interval, Above Normal | 0 | 1 | 0 | 0 | 1
  PR interval, Below Normal | 0 | 0 | 0 | 0 | 0
  PR interval, Within Normal | 10 | 9 | 10 | 10 | 9
  QTcB, Above Normal | 0 | 1 | 2 | 0 | 1
  QTcB, Below Normal | 0 | 0 | 0 | 0 | 0
  QTcB, Within Normal | 10 | 9 | 8 | 10 | 9
  QTcF, Above Normal | 1 | 0 | 1 | 0 | 2
  QTcF, Below Normal | 0 | 0 | 0 | 0 | 0
  QTcF, Within Normal | 9 | 10 | 9 | 10 | 8

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Laboratory parameters included hematology, clinical chemistry and urine parameters. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Any abnormal laboratory test results which were considered clinically significant by the investigator were recorded on the case report form. Number of participants with any clinically significant abnormalities in laboratory parameters have been presented.
Time Frame: Up to 50 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of BMS-626529 Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess Cmax of BMS-626529 following Q12H dosing. Geometric mean and geometric coefficient of variation are presented for Day 1, Day 8 morning dose (Anti Meridiem [AM]), Day 8 evening dose (Post Meridiem [PM]) and Day 8 morning + evening dose (AM+PM). Pharmacokinetic parameter values were derived by non-compartmental methods. Pharmacokinetic (PK) Population was used which comprised of all participants who receive BMS-663068 and provided pharmacokinetic samples.
Time Frame: Days 1, 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours
Population: PK Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10
Micrograms per milliliter (μg/mL)
  Day 1, n=10,10,10,10 | 1.74 (59.9) | 3.52 (26.6) | 4.05 (35.8) | 2.55 (27.4)
  Day 8, AM, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 8, AM, n=9,10,10,10 | 2.22 (67.1) | 5.55 (37.5) | 5.10 (57.4) | 3.18 (22.0)
  Day 8, PM, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 8, PM, n=9,10,10,10 | 2.25 (46.4) | 4.60 (29.2) | 4.77 (36.2) | 3.61 (27.5)
  Day 8, AM+PM, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 8, AM+PM, n=9,10,10,10 | 2.24 (43.3) | 5.05 (31.7) | 4.93 (40.1) | 3.39 (15.9)

11. Secondary Outcome: Cmax of BMS-626529 Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess Cmax of BMS-626529 following QHS dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1, Day 8 evening dose (PM) and Day 8 morning (AM) + evening dose (PM).
Time Frame: Days 1, 8: pre-evening dose, 1,2,3,4,5,6,8 hours
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 10
μg/mL
  Day 1, n=10 | 3.85 (32.0)
  Day 8, PM, n=9: number analyzed (Participants) | 9
  Day 8, PM, n=9 | 3.47 (31.7)
  Day 8, AM+PM, n=9: number analyzed (Participants) | 9
  Day 8, AM+PM, n=9 | 3.47 (31.7)

12. Secondary Outcome: Trough Observed Plasma Concentration (Ctrough) of BMS-626529 Following Q12H Dosing
Description: Blood samples were collected at indicated time points to access Ctrough of BMS-626529 following Q12H dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1, Days 5, 6, 7, 8, Day 8 morning dose (AM) and Day 8 evening dose (PM).
Time Frame: Days 1, 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours; Days 5,6,7: pre-morning dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10
Micrograms per milliliter (μg/mL)
  Day 1, n=10,10,10,10 | 0.349 (156) | 0.499 (83.4) | 0.640 (114) | 0.244 (78.3)
  Day 5, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 5, n=9,10,10,10 | 0.473 (119) | 1.04 (72.2) | 0.760 (67.1) | 0.518 (48.2)
  Day 6, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 6, n=9,10,10,10 | 0.436 (89.5) | 0.839 (49.1) | 0.737 (73.2) | 0.451 (49.2)
  Day 7, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 7, n=9,10,10,10 | 0.495 (96.5) | 1.08 (72.9) | 0.998 (91.8) | 0.542 (73.5)
  Day 8, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 8, n=9,10,10,10 | 0.460 (89.2) | 0.743 (47.1) | 0.720 (83.5) | 0.628 (76.9)
  Day 8, AM, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 8, AM, n=9,10,10,10 | 0.422 (69.1) | 0.951 (88.2) | 0.579 (71.5) | 0.469 (122)
  Day 8, PM, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 8, PM, n=9,10,10,10 | 0.358 (102) | 0.653 (109) | 0.553 (68.1) | 0.487 (47.5)

13. Secondary Outcome: Ctrough of BMS-626529 Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess Ctrough of BMS-626529 following QHS dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1, Days 5, 6, 7, 8 and Day 8 evening dose (PM).
Time Frame: Days 1, 8: pre-evening dose, 1,2,3,4,5,6,8 hours; Days 5,6,7: pre-evening dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 10
μg/mL
  Day 1, n=10 | 0.699 (93.4)
  Day 5, n=9: number analyzed (Participants) | 9
  Day 5, n=9 | 0.0705 (114)
  Day 6, n=9: number analyzed (Participants) | 9
  Day 6, n=9 | 0.0743 (97.7)
  Day 7, n=9: number analyzed (Participants) | 9
  Day 7, n=9 | 0.0719 (166)
  Day 8, n=9: number analyzed (Participants) | 9
  Day 8, n=9 | 0.0546 (146)
  Day 8, PM, n=9: number analyzed (Participants) | 9
  Day 8, PM, n=9 | 0.0544 (156)

14. Secondary Outcome: Area Under the Concentration-time Curve in One Dosing Interval (AUC [Tau]) of BMS-626529 Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess AUC (tau) of BMS-626529 following Q12H dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1, Day 8 morning dose (AM) and Day 8 evening dose (PM).
Time Frame: Days 1, 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10
Hour*micrograms per milliliter
  Day 1, n=10,10,10,10 | 9.16 (68.7) | 18.3 (28.8) | 20.6 (45.0) | 13.8 (28.3)
  Day 8, AM, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 8, AM, n=9,10,10,10 | 13.1 (62.7) | 29.9 (37.0) | 27.6 (48.4) | 19.5 (20.5)
  Day 8, PM, n=9,10,10,10: number analyzed (Participants) | 9 | 10 | 10 | 10
  Day 8, PM, n=9,10,10,10 | 13.1 (63.8) | 30.6 (26.3) | 27.0 (45.2) | 22.5 (34.0)

15. Secondary Outcome: AUC (Tau) of BMS-626529 Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess AUC (tau) of BMS-626529 following QHS dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1 and Day 8 evening dose (PM).
Time Frame: Days 1, 8: pre-evening dose, 1,2,3,4,5,6,8 hours
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 10
Hour*micrograms per milliliter
  Day 1, n=10 | 25.5 (38.0)
  Day 8 PM, n=9: number analyzed (Participants) | 9
  Day 8 PM, n=9 | 23.0 (48.2)

16. Secondary Outcome: Area Under the Concentration-time Curve Over a 24-hour Period (AUC [0-24]) of BMS-626529 Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess AUC (0-24) of BMS-626529 following Q12H dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 8.
Time Frame: Day 8: pre-morning dose, 1,2,3,4,5,6,8,12, 13,14,15,16,17,18,20 hours
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 10 | 10 | 10 | 10
Hour*micrograms per milliliter | 26.8 (56.1) | 60.6 (30.6) | 55.1 (44.3) | 42.6 (21.5)

17. Secondary Outcome: AUC (0-24) of BMS-626529 Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess AUC (0-24) of BMS-626529 following QHS dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 8.
Time Frame: Day 8: pre-evening dose, 1,2,3,4,5,6,8 hours
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 10
Hour*micrograms per milliliter | 23.0 (48.2)

18. Secondary Outcome: Accumulation Index (AI) of BMS-626529 Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess Accumulation Index of BMS-626529 following Q12H dosing. AI was calculated as ratio of AUC(tau) at steady-state to AUC(tau) after the first dose. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 8 morning dose (AM).
Time Frame: Day 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 9 | 10 | 10 | 10
Ratio of AUC | 1.53 (49.4) | 1.63 (26.7) | 1.34 (25.4) | 1.42 (37.0)

19. Secondary Outcome: Accumulation Index of BMS-626529 Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess Accumulation Index of BMS-626529 following QHS dosing. AI was calculated as ratio of AUC(tau) at steady-state to AUC(tau) after the first dose. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 8 evening dose (PM).
Time Frame: Day 8: pre-evening dose, 1,2,3,4,5,6,8 hours
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 9
Ratio of AUC | 0.912 (27.1)

20. Secondary Outcome: Inhibitory Quotient (IQ) of BMS-626529 by Css,Avg and by Lowest Concentration of a Drug During Dosing Interval (Cmin) Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess IQ of BMS-626529. Inhibitory quotient was calculated as the ratio of BMS-626529 in vivo exposure to in vitro measured protein binding adjusted EC90 (PBA-EC90). The following in vivo exposure measures were used in evaluating IQ: Cmin and Css,avg. Geometric mean and geometric coefficient of variation are presented.
Time Frame: Days 1, 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours; Day 9: pre-dose, 4,12 hours; Day 10: pre-dose, 12 hours; Day 11: pre-dose; Days 5,6,7: pre-morning dose
Population: PK Population. Only those participants with data available at the specified time points were analyzed. No evidence of a correlation between changes in viral load from Baseline (on Day 9 or the nadir) and the BMS-626529 PK parameters was found. Log10 PBA EC90 and IQs of Cmin and Css,avg were found to correlate with antiviral activity.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 8 | 9 | 10 | 10
Ratio
  IQ Cmin | 11.0 (3510) | 97.5 (382) | 67.2 (543) | 4.54 (21600)
  IQ Css,avg | 29.7 (4040) | 327 (454) | 252 (789) | 15.4 (14900)

21. Secondary Outcome: Inhibitory Quotient (IQ) of BMS-626529 by Css,Avg and by Lowest Concentration of a Drug During Dosing Interval (Cmin) Following QHS Dosing
Description: as for outcome 20
Time Frame: Days 1, 8: pre-evening dose, 1,2,3,4,5,6,8 hours; Day 2: pre-evening dose, 12,16 hours; Day 9: pre-dose, 12,16 hours; Day 10: pre-dose, 12 hours; Day 11: pre-dose; Days 5,6,7: pre-evening dose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 9
Ratio
  IQ Cmin | 3.86 (1070)
  IQ Css,avg | 67.8 (902)

22. Secondary Outcome: Inhibitory Quotient of BMS-626529 by Ctrough Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess IQ of BMS-626529. Inhibitory quotient was calculated as the ratio of BMS-626529 in vivo exposure to in vitro measured protein binding adjusted EC90 (PBA-EC90). The following in vivo exposure measure was used in evaluating IQ: Ctrough. Geometric mean and geometric coefficient of variation are presented.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
Number analyzed (Participants) | 8 | 9 | 10 | 10
Ratio | 12.2 (2750) | 120 (568) | 87.3 (763) | 4.61 (19000)

23. Secondary Outcome: Inhibitory Quotient of BMS-626529 by Ctrough Following QHS Dosing
Description: as for outcome 22
Time Frame: Days 1, 8: pre-evening dose, 1,2,3,4,5,6,8 hours; Days 2: pre-evening dose, 12,16 hours; Day 9: pre-dose, 12,16 hours; Day 10: pre-dose, 12 hours; Day 11: pre-dose; Days 5,6,7: pre-evening dose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 9
Ratio | 4.77 (1010)

24. Secondary Outcome: Cmax of Ritonavir Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess Cmax of ritonavir following Q12H dosing. Geometric mean and geometric coefficient of variation are presented for Day 1, Day 8 morning dose (AM), Day 8 evening dose (PM) and Day 8 morning + evening dose (AM+PM). Pharmacokinetic parameter values were derived by non-compartmental methods. PK Population was used which comprised of all participants who receive ritonavir and provided pharmacokinetic samples.
Time Frame: Days 1, 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM
Number analyzed (Participants) | 10 | 10 | 10
Micrograms per milliliter (μg/mL)
  Day 1, n=10,10,10 | 0.330 (91.3) | 0.314 (111) | 0.294 (59.6)
  Day 8, AM, n=9,10,10: number analyzed (Participants) | 9 | 10 | 10
  Day 8, AM, n=9,10,10 | 1.31 (101) | 1.30 (58.3) | 0.841 (44.9)
  Day 8, PM, n=9,10,0: number analyzed (Participants) | 9 | 10 | 0
  Day 8, PM, n=9,10,0 | 1.24 (73.4) | 1.48 (47.7) |
  Day 8, AM+PM, n=9,10,10: number analyzed (Participants) | 9 | 10 | 10
  Day 8, AM+PM, n=9,10,10 | 1.27 (80.0) | 1.39 (50.7) | 0.841 (44.9)

25. Secondary Outcome: Cmax of Ritonavir Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess Cmax of ritonavir following QHS dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1, Day 8 evening dose (PM) and Day 8 morning (AM) + evening dose (PM).
Time Frame: Days 1, 8: pre-evening dose, 1,2,3,4,5,6,8 hours
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 10
μg/mL
  Day 1, n=10 | 0.257 (53.8)
  Day 8, PM, n=9: number analyzed (Participants) | 9
  Day 8, PM, n=9 | 0.628 (56.4)
  Day 8, AM+PM, n=9: number analyzed (Participants) | 9
  Day 8, AM+PM, n=9 | 0.628 (56.4)

26. Secondary Outcome: Ctrough of Ritonavir Following Q12H Dosing
Description: Blood samples were collected at indicated time points to access Ctrough of ritonavir following Q12H dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1, Days 5, 6, 7, 8, Day 8 morning dose (AM) and Day 8 evening dose (PM).
Time Frame: Days 1, 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours; Days 5,6,7: pre-morning dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM
Number analyzed (Participants) | 10 | 10 | 10
Micrograms per milliliter (μg/mL)
  Day 1, n=10,10,0: number analyzed (Participants) | 10 | 10 | 0
  Day 1, n=10,10,0 | 0.117 (90.1) | 0.131 (98.2) |
  Day 5, n=9,10,10: number analyzed (Participants) | 9 | 10 | 10
  Day 5, n=9,10,10 | 0.502 (84.3) | 0.554 (73.9) | 0.0831 (77.8)
  Day 6, n=9,10,10: number analyzed (Participants) | 9 | 10 | 10
  Day 6, n=9,10,10 | 0.526 (87.9) | 0.594 (77.0) | 0.0820 (77.9)
  Day 7, n=9,10,10: number analyzed (Participants) | 9 | 10 | 10
  Day 7, n=9,10,10 | 0.477 (93.5) | 0.587 (76.3) | 0.0860 (79.9)
  Day 8, n=9,10,10: number analyzed (Participants) | 9 | 10 | 10
  Day 8, n=9,10,10 | 0.470 (90.6) | 0.503 (73.2) | 0.0891 (81.7)
  Day 8, AM, n=9,10,10: number analyzed (Participants) | 9 | 10 | 10
  Day 8, AM, n=9,10,10 | 0.345 (105) | 0.393 (66.3) | 0.0912 (70.5)
  Day 8, PM, n=9,10,0: number analyzed (Participants) | 9 | 10 | 0
  Day 8, PM, n=9,10,0 | 0.453 (86.2) | 0.476 (77.9) |

27. Secondary Outcome: Ctrough of Ritonavir Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess Ctrough of ritonavir following QHS dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1, Days 5, 6, 7, 8 and Day 8 evening dose (PM).
Time Frame: Days 1, 8: pre-evening dose, 1,2,3,4,5,6,8 hours; Days 5,6,7: pre-evening dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 10
μg/mL
  Day 1, n=10 | 0.157 (87.0)
  Day 5, n=9: number analyzed (Participants) | 9
  Day 5, n=9 | 0.107 (69.4)
  Day 6, n=9: number analyzed (Participants) | 9
  Day 6, n=9 | 0.0845 (67.7)
  Day 7, n=9: number analyzed (Participants) | 9
  Day 7, n=9 | 0.0844 (65.0)
  Day 8, n=9: number analyzed (Participants) | 9
  Day 8, n=9 | 0.0808 (73.2)
  Day 8, PM, n=9: number analyzed (Participants) | 9
  Day 8, PM, n=9 | 0.0830 (71.7)

28. Secondary Outcome: AUC (Tau) of Ritonavir Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess AUC (tau) of ritonavir following Q12H dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1, Day 8 morning dose (AM) and Day 8 evening dose (PM).
Time Frame: Days 1, 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM
Number analyzed (Participants) | 10 | 10 | 10
Hour*micrograms per milliliter
  Day 1, n=10,10,0: number analyzed (Participants) | 10 | 10 | 0
  Day 1, n=10,10,0 | 2.37 (99.5) | 2.05 (104) |
  Day 8, AM, n=9,10,10: number analyzed (Participants) | 9 | 10 | 10
  Day 8, AM, n=9,10,10 | 9.43 (89.1) | 9.05 (62.8) | 6.76 (49.3)
  Day 8, PM, n=9,10,0: number analyzed (Participants) | 9 | 10 | 0
  Day 8, PM, n=9,10,0 | 9.23 (77.1) | 10.4 (52.4) |

29. Secondary Outcome: AUC (Tau) of Ritonavir Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess AUC (tau) of ritonavir following QHS dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 1 and Day 8 evening dose (PM).
Time Frame: Days 1, 8: pre-evening dose, 1,2,3,4,5,6,8 hours
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 10
Hour*micrograms per milliliter
  Day 1, n=10 | 2.91 (80.4)
  Day 8 PM, n=9: number analyzed (Participants) | 9
  Day 8 PM, n=9 | 6.13 (94.3)

30. Secondary Outcome: AUC (0-24) of Ritonavir Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess AUC (0-24) of ritonavir following Q12H dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 8.
Time Frame: Day 8: pre-morning dose, 1,2,3,4,5,6,8,12, 13,14,15,16,17,18,20 hours
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM
Number analyzed (Participants) | 9 | 10 | 10
Hour*micrograms per milliliter | 18.9 (80.0) | 19.5 (56.6) | 6.76 (49.3)

31. Secondary Outcome: AUC (0-24) of Ritonavir Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess AUC (0-24) of ritonavir following QHS dosing. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 8.
Time Frame: Day 8: pre-evening dose, 1,2,3,4,5,6,8 hours
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 9
Hour*micrograms per milliliter | 6.13 (94.3)

32. Secondary Outcome: Accumulation Index of Ritonavir Following Q12H Dosing
Description: Blood samples were collected at indicated time points to assess Accumulation Index of ritonavir following Q12H dosing. AI was calculated as ratio of AUC(tau) at steady-state to AUC(tau) after the first dose. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 8 morning dose (AM).
Time Frame: Day 8: pre-morning dose, 1,2,3,4,5,6,8,12 hours; Day 8: 13,14,15,16,17,18,20 hours
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM
Number analyzed (Participants) | 9 | 10 | 10
Ratio of AUC | 3.58 (64.0) | 4.41 (41.7) | 3.62 (39.8)

33. Secondary Outcome: Accumulation Index of Ritonavir Following QHS Dosing
Description: Blood samples were collected at indicated time points to assess Accumulation Index of ritonavir following QHS dosing. AI was calculated as ratio of AUC(tau) at steady-state to AUC(tau) after the first dose. Pharmacokinetic parameter values were derived by non-compartmental methods. Geometric mean and geometric coefficient of variation are presented for Day 8 evening dose (PM).
Time Frame: Day 8: pre-evening dose, 1,2,3,4,5,6,8 hours
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | BMS-663068 1200 mg QHS + RTV 100 mg QHS
Number analyzed (Participants) | 9
Ratio of AUC | 2.19 (16.2)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and Non-serious adverse events (Non-SAEs) were collected from the start of the study treatment up to 50 days.
Description: SAEs and Non-SAEs were reported by treatment for the Safety Population which comprised of all randomized participants who used the trial medication at least once.
Arm/Group | BMS-663068 600 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg QHS + RTV 100 mg QHS | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H | BMS-663068 1200 mg Q12H + RTV 100 mg QAM | BMS-663068 1200 mg Q12H
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 5/10 | 9/10 | 8/10 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-663068 600 mg Q12H + RTV 100 mg Q12H (N=10) | BMS-663068 1200 mg QHS + RTV 100 mg QHS (N=10) | BMS-663068 1200 mg Q12H + RTV 100 mg Q12H (N=10) | BMS-663068 1200 mg Q12H + RTV 100 mg QAM (N=10) | BMS-663068 1200 mg Q12H (N=10)
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
EYE PRURITUS (Eye disorders) | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 1
DISCOMFORT (General disorders) | 0 | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 1 | 0 | 1 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 0 | 0 | 0
ABSCESS JAW (Infections and infestations) | 0 | 0 | 1 | 0 | 0
GONORRHOEA (Infections and infestations) | 0 | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 3 | 2 | 0
RHINITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 4 | 3 | 4 | 3 | 4
NEURALGIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
DISORIENTATION (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2
LISTLESS (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 1 | 1 | 1 | 1 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1 | 2
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2010-03-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT01009814/Prot_000.pdf
  • Statistical Analysis Plan (2010-09-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT01009814/SAP_001.pdf